CLINICAL TRIAL: NCT01661907
Title: Effects of Two Different Anesthesia-analgesia Methods on the Incidence of Postoperative Delirium: a Multicenter, Randomized Controlled Trial
Brief Title: Anesthesia-analgesia Methods and Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Peking University Third Hospital (Other); Beijing Hospital (Other Government); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PUCRP201101; ChiCTR-TRC-09000543 (Registry Identifier: Chinese Clinical Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Elderly; Epidural Anesthesia; General Anesthesia; Major Surgery; Postoperative Delirium
Keywords: Elderly; Epidural anesthesia; General anesthesia; Major surgery; Postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Epi-GA/PCEA (Experimental): Patients assigned to this group (experimental group) will receive combined epidural-general anesthesia (combined Epi-GA) and patient-controlled epidural analgesia (PCEA).
  An epidural catheter will be placed before anesthesia induction. General anesthesia will be induced and maintained in the same manner as in the control group, with the addition of a continuous infusion or intermittent boluses of 0.375%-0.5% ropivacaine given through the epidural catheter for analgesia maintenance. Patient-controlled epidural analgesia will be provided for postoperative analgesia (established with 0.12% ropivacaine and 0.5 μg/mL sufentanil in 250 mL normal saline, programmed to deliver a 2-mL bolus with a lockout interval of 20 minutes and a background infusion of 4 mL/hr).
  Interventions: Procedure: Combined Epi-GA/PCEA
- GA/PCIA (Active Comparator): Patients assigned to this group (control group) will receive general anesthesia (GA) and patient-controlled intravenous analgesia (PCIA).
  General anesthesia will be induced with midazolam, sufentanil, propofol and rocuronium. Anesthesia will then be maintained by inhalation of sevoflurane with or without nitrous oxide, and/or continuous intravenous infusion of propofol. Sufentanil and rocuronium will be given when needed. Patient-controlled intravenous analgesia will be provided for postoperative analgesia (established with 50 mg morphine in 100 mL normal saline, programmed to deliver a 2-mL bolus with a 6-10 minutes lockout interval and a 1 mL/hr background infusion).
  Interventions: Procedure: GA/PCIA

INTERVENTIONS:
Procedure: Combined Epi-GA/PCEA — An epidural catheter will be placed before the induction of general anesthesia. General anesthesia will be induced and maintained as in the control group, with the addition of epidural anesthesia which will be maintained with the use of 0.375%-0.5% ropivacaine during surgery. Patient-controlled epidural analgesia will be provided after surgery.
  Arms: Combined Epi-GA/PCEA
Procedure: GA/PCIA — General anesthesia will be induced with midazolam, propofol, sufentanil and rocuronium. Anesthesia will be maintained with either intravenous (propofol), inhalational (sevoflurane with or without nitrous oxide), or combined intravenous-inhalational anesthetics. Additional opioids (remifentanil, sufentanil, fentanyl, or morphine) and muscle relaxant (rocuronium, atracurium, or cisatracurium) will be administered when deemed necessary by the attending anesthesiologists. Patient-controlled intravenous analgesia will be provided after surgery.
  Arms: GA/PCIA

SUMMARY:
Postoperative delirium is a common complication in elderly patients after surgery. Its occurrence is associated with worse outcomes. The pathophysiology of delirium remains poorly understood. However, an universal phenomenon is that delirium frequently occurs in elderly patients after major complicated surgery, but is rarely seen after minor ambulatory surgery (such as cataract surgery). This indicates that stress response produced by surgery might have an important role in the pathogenesis of delirium. It has been reported that, when compared with general anesthesia and postoperative intravenous analgesia, neuraxial anesthesia and analgesia reduced the occurrence of postoperative complications and mortality in high risk patients. Combined epidural-general anesthesia is frequently used in clinical practice. This anesthetic method provides advantages of both epidural and general anesthesia, i.e. it blocks the afferent pathway of nociceptive stimulus by neuraxial blockade during and after surgery, and allows patients to endure long-duration surgery without any awareness. The investigators hypothesize that combined epidural-general anesthesia and postoperative epidural analgesia can decrease the incidence of delirium in elderly patients after major surgery when compared with general anesthesia alone and postoperative intravenous analgesia.

DETAILED DESCRIPTION:
Delirium is an acutely occurred and transient mental syndrome characterized by global impairment of cognitive functions, reduced level of consciousness, abnormalities of attention, increased or decreased psychomotor activity, and disordered sleep-wake cycle. Postoperative delirium is a common complication in elderly patients after surgery. Dyer et al reviewed 80 primary studies and found that the mean incidence of postoperative delirium is about 36.8% (range 0%-73.5%) after surgery. It occurs in up to 80% of patients in the intensive care unit (ICU). Our recent studies found that delirium occurred in 51.0% of patients after cardiac surgery and in 44.5% of patients after non-cardiac surgery.

The occurrence of postoperative delirium is associated with worse outcomes. Studies showed that delirious patients have prolonged ICU stay, increased incidence of complications, prolonged hospitalization, high mortality rate, and increased health care costs. Delirium is also associated with increased risk of long-term cognitive decline and poor quality of life. A recent follow-up study (mean follow-up time 27.9 ± 3.1 months) by our research group found that, after adjusting factors such as age, occurrence of postoperative complications, and stage of cancer, etc, the occurrence of postoperative delirium still remained an independent predictor of long-term mortality.

The pathophysiology of delirium remains poorly understood. An universal phenomenon is that delirium frequently occurs in elderly patients after major complicated surgery, but is rarely seen after minor ambulatory surgery (such as cataract surgery). Studies also found that postoperative pain is an independent risk factor of delirium, whereas effective pain relief may help to reduce the incidence of delirium. Our recent studies showed that high serum cortisol level is an independent risk factor of postoperative delirium. In addition, inflammatory response may also contribute to the pathogenesis of delirium. Trauma, pain, cortisol secretion and inflammation are all important components of surgical stress response. The above results indicated that stress response produced by surgery might have an important role in the pathogenesis of delirium.

Previous studies demonstrated that, when compared with general anesthesia, neuraxial anesthesia attenuates the hypersecretion of cortisol, and decreases the intensity of inflammatory response more effectively after surgery. And epidural analgesia provides better postoperative pain relief than intravenous analgesia. It was also reported that, when compared with general anesthesia and intravenous analgesia, neuraxial anesthesia and analgesia reduces the occurrence of postoperative complications and mortality in high risk patients. Combined epidural-general anesthesia is frequently used in clinical practice, and is performed in about 1/4 of patients undergoing surgery in the applicant's hospital. Theoretically, this anesthetic method provides advantages of both epidural and general anesthesia, i.e. it blocks the afferent pathway of nociceptive stimulus by neuraxial blockade during and after surgery, and allow patients to endure long-duration complicated surgeries without any awareness. However, there is no evidence whether combined epidural-general anesthesia/postoperative epidural analgesia can decrease the incidence of postoperative delirium in elderly patients undergoing major surgery.

The objective of the study is to compare the effects of combined epidural-general anesthesia/postoperative epidural analgesia and general anesthesia/postoperative intravenous analgesia on the incidence of postoperative delirium in elderly patients undergoing major noncardiac surgery.

ELIGIBILITY:
Inclusion criteria:

1. elderly patients (age range 60-90 years);
2. scheduled to undergo noncardiac thoracic or abdominal surgery with an expected duration of 2 hours or longer. For those who undergo thoracoscopic or laparoscopic surgery, the expected length of incision must be 5 centimeters or more;
3. agree to receive patient-controlled postoperative analgesia.

Exclusion criteria (patients who meet any of the following criteria will be excluded):

1. previous history of schizophrenia, epilepsy or Parkinson disease, or unable to complete preoperative assessment due to severe dementia, language barrier or end-stage disease;
2. history of myocardial infarction within 3 months before surgery;
3. any contraindication to epidural anesthesia and analgesia, including abnormal vertebral anatomy, previous spinal trauma or surgery, severe chronic back pain, coagulation disorder (prothrombin time or activated partial prothrombin time longer than 1.5 times of the upper limit of normal, or platelet count of less than 80 × 10^9/L), local infection near the site of puncture, and severe sepsis;
4. severe heart dysfunction (New York Heart Association functional classification 3 or above), hepatic insufficiency (Child-Pugh grades C), or renal insufficiency (serum creatinine of 442 μmol/L or above, with or without serum potassium of 6.5 mmol/L or above, or requirement of renal replacement therapy); or
5. any other conditions that were considered unsuitable for study participation.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2015-05-25 (Actual); Study Completion 2015-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | During the first 7 days after surgery.
  Patients will be visited twice daily during the first seven days after surgery (between 08:00 h and 10:00 h, and between 18:00 h and 20:00 h). Delirium will be assessed with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). The incidence is calculated as percentage of patients who develope any episode of delirium during that period.

SECONDARY OUTCOMES:
Intensive care unit (ICU) admission after surgery | During the day of surgery.
  The proportion of patients admitted to the ICU after surgery
APACHE II score at ICU admission | Within 24 hours after surgery.
  For patients admitted to the ICU after surgery, the worst Acute Physiology and Chronic Health Evaluation II (APACHE II) score within 24 h will be recorded.
The percentage of ICU admission with endotracheal intubation | During the day of surgery.
  The percentage of ICU admission with endotracheal intubation.
The duration of Mechanical Ventilation in ICU | Up to 30 days after surgery.
  For patients admitted to the ICU after surgery, the duration of mechanical ventilation (for those with endotracheal tubes) will be recorded.
The Length of ICU stay | Up to 30 days after surgery.
  For patients admitted to the ICU after surgery, the length of ICU stay will be recorded.
Time to the first onset of delirium | Up to 7 days after surgery.
  Patients will be visited twice daily during the first seven days after surgery (between 08:00 h and 10:00 h, and between 18:00 h and 20:00 h). Delirium will be assessed with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).
Time to fluid/food intake | Up to 30 days after surgery.
  Patients will be followed-up until 30 days after surgery and time to fluid and food intake after surgery will be recorded.
Length of stay in hospital after surgery | Up to 30 days after surgery.
  Patients will be followed-up until 30 days after surgery.
All-cause 30-day mortality | Within the first 30 days after surgery.
  All-cause 30-day mortality
Non-delirium complications within 30 days after surgery surgery | Within the first 30 days after surgery.
  Defined as newly occurred medical conditions other than delirium that are harmful to patients' postoperative recovery and required therapeutic intervention (i.e., grade II or higher on the Clavien-Dindo classification).
The intensity of postoperative pain | During the first 3 postoperative days.
  The intensity of postoperative pain both at rest and with movement will be evaluated twice daily at the same time of delirium assessment (between 08:00 h and 10:00 h, and between 18:00 h and 20:00 h) with the numeric rating scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain).

OTHER OUTCOMES:
Serum cortisol concentration (substudy) | Blood samples will be collected from selected patients before surgery, and in the morning of the 1st and 3rd day after surgery.
  Serum cortisol concentration (substudy)
Serum IL-6 concentration (substudy) | Blood samples will be collected from selected patients before surgery, and in the morning of the 1st and 3rd day after surgery.
  Serum IL-6 concentration (substudy)
Serum IL-8 concentration (substudy) | Blood samples will be collected from selected patients before surgery, and in the morning of the 1st and 3rd day after surgery.
  Serum IL-8 concentration (substudy)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hopital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data will be provided on request.

REFERENCES:
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Mu DL, Wang DX, Li LH, Shan GJ, Li J, Yu QJ, Shi CX. High serum cortisol level is associated with increased risk of delirium after coronary artery bypass graft surgery: a prospective cohort study. Crit Care. 2010;14(6):R238. doi: 10.1186/cc9393. Epub 2010 Dec 30. PMID 21192800
- [Background] Shi CM, Wang DX, Chen KS, Gu XE. Incidence and risk factors of delirium in critically ill patients after non-cardiac surgery. Chin Med J (Engl). 2010 Apr 20;123(8):993-9. PMID 20497703
- [Background] Roberts B, Rickard CM, Rajbhandari D, Turner G, Clarke J, Hill D, Tauschke C, Chaboyer W, Parsons R. Multicentre study of delirium in ICU patients using a simple screening tool. Aust Crit Care. 2005 Feb;18(1):6, 8-9, 11-4 passim. doi: 10.1016/s1036-7314(05)80019-0. PMID 18038529
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Milstein A, Pollack A, Kleinman G, Barak Y. Confusion/delirium following cataract surgery: an incidence study of 1-year duration. Int Psychogeriatr. 2002 Sep;14(3):301-6. doi: 10.1017/s1041610202008499. PMID 12475090
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Hudek K. Emergence delirium: a nursing perspective. AORN J. 2009 Mar;89(3):509-16; quiz 517-9. doi: 10.1016/j.aorn.2008.12.026. PMID 19326585
- [Background] Rudolph JL, Ramlawi B, Kuchel GA, McElhaney JE, Xie D, Sellke FW, Khabbaz K, Levkoff SE, Marcantonio ER. Chemokines are associated with delirium after cardiac surgery. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):184-9. doi: 10.1093/gerona/63.2.184. PMID 18314455
- [Background] de Rooij SE, van Munster BC, Korevaar JC, Levi M. Cytokines and acute phase response in delirium. J Psychosom Res. 2007 May;62(5):521-5. doi: 10.1016/j.jpsychores.2006.11.013. PMID 17467406
- [Background] van Munster BC, Korevaar JC, Zwinderman AH, Levi M, Wiersinga WJ, De Rooij SE. Time-course of cytokines during delirium in elderly patients with hip fractures. J Am Geriatr Soc. 2008 Sep;56(9):1704-9. doi: 10.1111/j.1532-5415.2008.01851.x. Epub 2008 Aug 4. PMID 18691278
- [Background] Li Y, Zhu S, Yan M. Combined general/epidural anesthesia (ropivacaine 0.375%) versus general anesthesia for upper abdominal surgery. Anesth Analg. 2008 May;106(5):1562-5, table of contents. doi: 10.1213/ane.0b013e31816d1976. PMID 18420877
- [Background] Ahlers O, Nachtigall I, Lenze J, Goldmann A, Schulte E, Hohne C, Fritz G, Keh D. Intraoperative thoracic epidural anaesthesia attenuates stress-induced immunosuppression in patients undergoing major abdominal surgery. Br J Anaesth. 2008 Dec;101(6):781-7. doi: 10.1093/bja/aen287. Epub 2008 Oct 15. PMID 18922851
- [Background] Pham-Marcou TA, Gentili M, Asehnoune K, Fletcher D, Mazoit JX. Effect of neurolytic nerve block on systemic carrageenan-induced inflammatory response in mice. Br J Anaesth. 2005 Aug;95(2):243-6. doi: 10.1093/bja/aei150. Epub 2005 Apr 29. PMID 15863437
- [Background] Behera BK, Puri GD, Ghai B. Patient-controlled epidural analgesia with fentanyl and bupivacaine provides better analgesia than intravenous morphine patient-controlled analgesia for early thoracotomy pain. J Postgrad Med. 2008 Apr-Jun;54(2):86-90. doi: 10.4103/0022-3859.40772. PMID 18480522
- [Background] Pisani MA, Murphy TE, Araujo KL, Slattum P, Van Ness PH, Inouye SK. Benzodiazepine and opioid use and the duration of intensive care unit delirium in an older population. Crit Care Med. 2009 Jan;37(1):177-83. doi: 10.1097/CCM.0b013e318192fcf9. PMID 19050611
- [Background] Saeki H, Ishimura H, Higashi H, Kitagawa D, Tanaka J, Maruyama R, Katoh H, Shimazoe H, Yamauchi K, Ayabe H, Kakeji Y, Morita M, Maehara Y. Postoperative management using intensive patient-controlled epidural analgesia and early rehabilitation after an esophagectomy. Surg Today. 2009;39(6):476-80. doi: 10.1007/s00595-008-3924-2. Epub 2009 May 27. PMID 19468802
- [Background] Ballantyne JC, Kupelnick B, McPeek B, Lau J. Does the evidence support the use of spinal and epidural anesthesia for surgery? J Clin Anesth. 2005 Aug;17(5):382-91. doi: 10.1016/j.jclinane.2004.10.005. PMID 16102692
- [Background] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Background] Park WY, Thompson JS, Lee KK. Effect of epidural anesthesia and analgesia on perioperative outcome: a randomized, controlled Veterans Affairs cooperative study. Ann Surg. 2001 Oct;234(4):560-9; discussion 569-71. doi: 10.1097/00000658-200110000-00015. PMID 11573049
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Bryson GL, Wyand A. Evidence-based clinical update: general anesthesia and the risk of delirium and postoperative cognitive dysfunction. Can J Anaesth. 2006 Jul;53(7):669-77. doi: 10.1007/BF03021625. PMID 16803914
- [Background] Kamitani K, Higuchi A, Asahi T, Yoshida H. [Postoperative delirium after general anesthesia vs. spinal anesthesia in geriatric patients]. Masui. 2003 Sep;52(9):972-5. Japanese. PMID 14531256
- [Background] Papaioannou A, Fraidakis O, Michaloudis D, Balalis C, Askitopoulou H. The impact of the type of anaesthesia on cognitive status and delirium during the first postoperative days in elderly patients. Eur J Anaesthesiol. 2005 Jul;22(7):492-9. doi: 10.1017/s0265021505000840. PMID 16045136
- [Derived] Li YW, Li HJ, Li HJ, Feng Y, Yu Y, Guo XY, Li Y, Zhao BJ, Hu XY, Zuo MZ, Zhang HY, Wang MR, Ji P, Yan XY, Wu YF, Wang DX. Effects of two different anesthesia-analgesia methods on incidence of postoperative delirium in elderly patients undergoing major thoracic and abdominal surgery: study rationale and protocol for a multicenter randomized controlled trial. BMC Anesthesiol. 2015 Oct 13;15:144. doi: 10.1186/s12871-015-0118-5. PMID 26459347